CLINICAL TRIAL: NCT01949922
Title: Treatment of Fecal Incontinence by Injection of Autologous Muscle Fibers Into the Anal Sphincter - a Pilot Study.
Brief Title: Treatment of Fecal Incontinence by Injection of Autologous Muscle Fibers Into the Anal Sphincter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Hanna Jangö, MD, PhD-student, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2013-027
Record Dates: First submitted 2013-04-11; First posted 2013-09-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Fecal Incontinence; Anal Incontinence
Keywords: regenerative medicine; fecal incontinence; muscle fiber injection
MeSH Terms: conditions — Fecal Incontinence; Encopresis | interventions — Diet Therapy; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injection of autologous muscle fibers in the anal sphincter (Experimental): All patients, that still have relevant symptoms after completion of three months with individualized pelvic floor muscle training and dietary intervention to control defecatory function, will be offered injection of autologous muscle fiber fragments in the anal sphincter. A myscle biopsy will be taken from the leg, cut into small pieces in a saline solution and injected in the anal sphincter.
  Interventions: Procedure: Injection of autologous muscle fibers into the anal sphincter.; Procedure: Pelvic floor muscle training; Behavioral: Dietary intervention; Drug: Analgesia

INTERVENTIONS:
Procedure: Injection of autologous muscle fibers into the anal sphincter.
Procedure: Pelvic floor muscle training — Pelvic floor muscle training 3 months to optimize pelvic floor muscle function. Autologous muscle stem cell injection will only be offered to patients that still have problems after completion of pelvic floor muscle training.
Behavioral: Dietary intervention — Dietary intervention 3 months to optimize defecatory function. Autologous muscle stem cell injection will only be offered to patients that still have problems after completion of pelvic floor muscle training and dietary intervention.
Drug: Analgesia — Patients will be offered analgesia as needed during and after surgery. Specific products will depend on allergy and preferences of doctors involved and patient's requirements.

SUMMARY:
Aim:

To investigate efficacy and safety in a new treatment with injection of autologous muscle fibers into the anal sphincter in patients with fecal incontinence.

Method:

Patients with fecal incontinence after obstetric anal sphincter rupture will be included. After inclusion, they will be offered 3 months of pelvic floor muscle training. If the patients after completion of pelvic floor muscle training still suffer from fecal incontinence, the patients will be offered treatment with autologous muscle fiber injection into the anal sphincter. The patients will be followed one year after the injection. The autologous muscle fibers are harvested at the patients leg muscle, cut into small pieces and injected into the anal sphincter. A small part of the fibers are used for analysing number of muscle stem cells and thereby the regenerative potential of the sample.

The study is a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* fecal incontinence
* Wexner score >= 9 or affected quality of life.
* Understanding and speaking danish
* Informed consent

Exclusion Criteria:

* Ongoing pregnancy
* Delivery in the last 12 months
* colostomy
* chronic inflammatory bowel disease (mb. crohn, colitis ulcerosa)
* improvement after pelvic floor muscle training in an extent that makes autologous muscle fiber injection unnecessary.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment using fecal incontinence score: Wexner score. | 1 year

SECONDARY OUTCOMES:
Safety | 1 year
  Number of adverse events, pain etc.

OTHER OUTCOMES:
Improvement of life quality | 1 year
Improvement of anal sphincter functioning assessed by anal reflectometry | 1 year.
Improvement of fecal incontinence after pelvic floor muscle training. | 3 months
Improvement of the anal sphincter by 3D ultrasound. | 1 year
Correlation between the tissue samples regenerative potential and effect of treatment. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Herlev University Hospital, Copenhagen, Herlev, Denmark